CLINICAL TRIAL: NCT00212615
Title: XELOX III. Capecitabine (Xeloda) in Combination With Oxaliplatin (Eloxatin) as First-line Treatment of Patients With Advanced or Metastatic Colorectal Cancer. A Randomized Phase II Study
Brief Title: XELOX III. Xeloda in Combination With Eloxatin for Patients With Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Per Pfeiffer, Professor, M.D., Odense University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: XELOX III; KFE 03.17
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: C04.588.274.476.411.307
Keywords: Colorectal neoplasm; Capecitabine (Xeloda); Oxaliplatin (Eloxatin); Advanced disease; Metastatic disease; First-line treatment; Phase II study
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Oxaliplatin; Capecitabine

ARMS (2):
- A (Active Comparator): Standard XELOX
  Interventions: Drug: Oxaliplatin (Eloxatin); Drug: Capecitabine (Xeloda)
- B (Active Comparator): Chronomodulated XELOX
  Interventions: Drug: Oxaliplatin (Eloxatin); Drug: Capecitabine (Xeloda)

INTERVENTIONS:
Drug: Oxaliplatin (Eloxatin)
Drug: Capecitabine (Xeloda)

SUMMARY:
XELOX (Capecitabine and Oxaliplatin) is an effective and convenient regimen for patients with metastatic colorectal cancer. Chronomodulated therapy may reduce toxicity. Patients will be randomized to standard XELOX (Capecitabine 1000 mg/m² in the morning and 1000 mg/m² in the evening days 1-14 and short term Oxaliplatin 130 mg/m² day 1 in 30 minutes) or chronomodulated XELOX (Capecitabine 400 mg/m² in the morning and 1600 mg/m² in the evening days 1-14 and short term Oxaliplatin 130 mg/m² day 1 in 30 minutes).

Bloodsamples will be collected and frozen and later examined for potential predictive factors

ELIGIBILITY:
Inclusion Criteria:

* Histological proven adenocarcinoma of the colon or rectum
* Measurable or non-measurable disease
* Performance status 0-2
* Adequate renal and hepatic functions
* Adjuvant chemotherapy must have ended 180 days before inclusion
* Written informed consent prior to randomization

Exclusion Criteria:

* Prior treatment with Eloxatin or Xeloda
* Peripheral neuropathy
* Evidence of CNS metastasis
* Other serious illness or medical conditions (including contraindication to 5 FU e.g.: angor, myocardial infarction within 6 months)
* Past history of malignant neoplasm within the past five years, except curatively treated non melanoma skin cancer
* Administration of any other experimental drug under investigation within 2 weeks before randomisation
* Pregnant or breast feeding women
* Fertile patients must use adequate contraceptives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2004-02 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Toxicity: before treatment (each 3 weeks) and by SAE (Serious Adverse Event)

SECONDARY OUTCOMES:
Physical examination: before treatment (each 3 weeks)
Performance status: before treatment (each 3 weeks)
Haematology: before treatment (each 3 weeks)
Tumor biology: after 1st treatment, every 9th weeks herafter
Biochemistry: after every 3rd treatment (each 9th weeks)
Tumor assesment: after every 3rd treatment (each 9th weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Per Pfeiffer, MD, Principal Investigator — Department of Oncology, Odense University Hospital
Locations (8):
- Denmark (6):
  - Department of Oncology, Esbjerg Hospital, Esbjerg
  - Department of Oncology, Herlev University Hospital, Herlev
  - Department of Oncology, Herning Hospital, Herning
  - Department of Oncology, Hillerød Hospital, Hillerød
  - Department of Oncology, Næstved Hospital, Næstved
  - Department of Oncology, Roskilde Hospital, Roskilde
- Sweden (2):
  - Department of Oncology, Radiumhemmet, Stockholm
  - Department of Oncology, Uppsala University Hospital, Uppsala

REFERENCES:
- [Background] Pfeiffer P, Hahn P, Jensen HA. Short-time infusion of oxaliplatin (Eloxatin) in combination with capecitabine (Xeloda) in patients with advanced colorectal cancer. Acta Oncol. 2003;42(8):832-6. doi: 10.1080/02841860310015894. PMID 14968944
- [Derived] Boisen MK, Johansen JS, Dehlendorff C, Larsen JS, Osterlind K, Hansen J, Nielsen SE, Pfeiffer P, Tarpgaard LS, Hollander NH, Keldsen N, Hansen TF, Jensen BB, Jensen BV. Primary tumor location and bevacizumab effectiveness in patients with metastatic colorectal cancer. Ann Oncol. 2013 Oct;24(10):2554-2559. doi: 10.1093/annonc/mdt253. Epub 2013 Jul 17. PMID 23864097